CLINICAL TRIAL: NCT03110133
Title: A Multicenter, Double-Blind, Parallel-Arm, Placebo-Controlled, Phase 2 Study of the Efficacy, Safety, and Tolerability of Oral Full-Spectrum MicrobiotaTM (CP101) in Subjects With Recurrence of Clostridium Difficile Infection
Brief Title: Efficacy, Safety, and Tolerability Study of Oral Full-Spectrum MicrobiotaTM (CP101) in Subjects With Recurrent C. Diff
Acronym: PRISM3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Finch Research and Development LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDI-001
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Clostridium Difficile Infection Recurrence
Keywords: Clostridium Difficile Infection; CP101; Crestovo; FMT; CDI; C. difficile; C. diff; Recurrent Clostridium Difficile Infection; Recurrent C. diff; Recurrent CDI; Finch; Fecal transplant; Fecal microbiota transplant; rCDI; Finch Therapeutics
MeSH Terms: conditions — Clostridium Infections; Diabetes Insipidus, Neurogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CP101 (Experimental): Full Spectrum Microbiota Capsule
  Interventions: Drug: Full Spectrum Microbiota
- Placebo (Placebo Comparator): Matching Placebo Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Full Spectrum Microbiota — Orally administered donor derived microbiota
  Other Names: CP101, FSM
  Arms: CP101
Drug: Placebo — Placebo for CP101
  Arms: Placebo

SUMMARY:
Subjects with recurrent C. difficile infection will receive an oral dose of CP101 capsules one time in Treatment Group I or matching placebo one time in Treatment Group II. The purpose of this study is to demonstrate the safety and effectiveness of CP101 to prevent recurrence of C. difficile.

Subjects with confirmed C. difficile recurrence within 8 weeks after administration of study drug (CP101 or placebo) may be eligible to enroll in the open-label extension study (CP101-CDI-E02) and will receive CP101.

DETAILED DESCRIPTION:
This is a Multicenter, Double-Blind, Parallel-Arm, Placebo-Controlled, Phase 2 Study of the Efficacy, Safety, and Tolerability of Oral Full-Spectrum MicrobiotaTM (CP101) in Subjects with Recurrence of Clostridium difficile Infection (CDI).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Men or women 18 years of age or older
* Current diagnosis of a recurrence of non-severe, non-complicated CDI
* Subject has a clinical response to standard-of-care CDI antibiotics for the most recent CDI episode

Exclusion Criteria:

* Pregnant, breast-feeding, or considering becoming pregnant during the study
* Prior history, evidence, or diagnosis of inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis)
* Any prior diagnosis of diarrhea-predominant irritable bowel syndrome
* Systemic chemotherapy or radiation for the treatment of cancer during the 60 days prior to consent or planned during the 8 weeks following Randomization
* Prior fecal transplant for any condition, regardless of route of administration in the last year or plans to undergo during the study
* Major intra-abdominal surgery within the past 60 days prior to Screening
* History of total colectomy/ileostomy or bariatric surgery
* Admitted to, or expected to be admitted to an intensive care unit for any medical reason. Note: Residents of long term care facilities are eligible study entry
* Planned hospitalization or invasive surgery during the study
* Severe acute illness unrelated to CDI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (51):
  - Scottsdale, Scottsdale, Arizona
  - Los Angeles, Los Angeles, California
  - Murrieta, Murrieta, California
  - Oakland, Oakland, California
  - San Diego, San Diego, California
  - San Francisco, San Francisco, California
  - Aurora, Aurora, Colorado
  - Bridgeport, Bridgeport, Connecticut
  - Hamden, Hamden, Connecticut
  - Washington DC, Washington D.C., District of Columbia
  - Jacksonville, Jacksonville, Florida
  - Naples, Naples, Florida
  - Pinellas Park, Pinellas Park, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Burr Ridge, Burr Ridge, Illinois
  - Chicago, Chicago, Illinois
  - Evanston, Evanston, Illinois
  - Maywood, Maywood, Illinois
  - Indianapolis, Indianapolis, Indiana
  - West Des Moines, West Des Moines, Iowa
  - Shawnee, Shawnee Mission, Kansas
  - New Orleans, New Orleans, Louisiana
  - Boston, Boston, Massachusetts
  - Detroit, Detroit, Michigan
  - Royal Oak, Royal Oak, Michigan
  - Rochester, Rochester, Minnesota
  - St. Paul, Saint Paul, Minnesota
  - Butte, Butte, Montana
  - Morristown, Morristown, New Jersey
  - Somers Point, Somers Point, New Jersey
  - New York, New York, New York
  - Bronx, The Bronx, New York
  - Chapel Hill, Chapel Hill, North Carolina
  - Kinston, Kinston, North Carolina
  - Pinehurst, Pinehurst, North Carolina
  - Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Poland, Poland, Ohio
  - Portland, Portland, Oregon
  - Lancaster, Lancaster, Pennsylvania
  - Providence, Providence, Rhode Island
  - Nashville, Nashville, Tennessee
  - San Antonio, San Antonio, Texas
  - Ogden, Ogden, Utah
  - Salt Lake City, Salt Lake City, Utah
  - Annandale, Annandale, Virginia
  - Charlottesville, Charlottesville, Virginia
  - Seattle, Seattle, Washington
  - Grafton, Grafton, Wisconsin
- Canada (3):
  - Calgary, Calgary, Alberta
  - Halifax, Halifax, Nova Scotia
  - Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allegretti JR, Kelly CR, Louie T, Fischer M, Hota S, Misra B, Van Hise NW, Yen E, Bullock JS, Silverman M, Davis I, McGill SK, Pardi DS, Orenstein R, Grinspan A, El-Nachef N, Feuerstadt P, Borody TJ, Khanna S, Budree S, Kassam Z. Safety and Tolerability of CP101, a Full-Spectrum, Oral Microbiome Therapeutic for the Prevention of Recurrent Clostridioides difficile Infection: A Phase 2 Randomized Controlled Trial. Gastroenterology. 2025 Feb;168(2):357-366.e3. doi: 10.1053/j.gastro.2024.09.030. Epub 2024 Oct 2. PMID 39366468

RESULTS

PARTICIPANT FLOW:
Period: Week 8
Arm/Group | CP101 | Placebo
Started | 106 | 100
Completed | 101 | 96
Not Completed | 5 | 4
Period: Week 24
Arm/Group | CP101 | Placebo
Started | 101 | 96
Completed | 99 | 95
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) population used
Groups:
- Total: Total of all reporting groups
Arm/Group | CP101 | Placebo | Total
Number analyzed (Participants) | 102 | 96 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (17.26) | 66.5 (14.25) | 66.2 (15.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 65 | 134
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 96 | 90 | 186
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 93 | 89 | 182
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 102 | 96 | 198
Total Number of C. difficile Infection (CDI) Episodes in Previous 12 Months [Count of Participants; unit: Participants]
  1 | 1 | 0 | 1
  2 | 37 | 29 | 66
  3 | 46 | 48 | 94
  >3 | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Recurrence Through Week 8 Based on Adjudication
Description: Defined in the protocol as sustained clinical cure
Time Frame: Week 8
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 102 | 96
Participants | 76 | 59
Statistical Analysis 1: Comparison: CP101 vs Placebo; Test type: Superiority; p = 0.0488, Chi-squared

2. Primary Outcome: Number of Participants With Occurrence of Treatment Emergent Adverse Events
Description: Mapped to System Organ Class. Any adverse event (AE) reported that occurs during or post the administration of IP is defined as a Treatment Emergent AE (TEAE)
Time Frame: Week 8
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 104 | 99
Participants | 96 | 88

3. Secondary Outcome: Time to First Recurrent CDI Episode During the Study
Description: The number of days between IP administration and the first C. Difficile recurrence
Time Frame: Week 8
Population: mITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 102 | 96
Days | 17.1 (10.95) | 11.3 (6.92)

4. Secondary Outcome: Number of Participants With Absence of Recurrence Through Week 24 Based on Adjudication
Description: Defined in the protocol as sustained clinical cure
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 102 | 96
Participants | 75 | 57
Statistical Analysis 1: Comparison: CP101 vs Placebo; Test type: Superiority; p = 0.0347, Chi-squared

5. Secondary Outcome: Number of Participants With Recurrence by Ribosomal NAP1/BI/027 C. Difficile Subtype
Description: NAP1 is the North American Pulse-field C. difficile subtype.
Time Frame: Up to Week 8
Population: Analysis population only included participants with a CDI recurrence up to week 8. Two of the recurrences in the primary efficacy analyses were imputed, therefore only 24 samples were available for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CP101 | Placebo
Number analyzed (Participants) | 24 | 37
Participants
  Ribosomal NAP1/BI/027 Positive at Recurrence | 6 | 7
  Ribosomal NAP1/BI/027 Negative or Unknown at Recurrence | 18 | 30

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Based on Safety population
Arm/Group | CP101 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/104 | 2/99
Serious Adverse Events (participants affected / at risk) | 16/104 | 13/99
Other Adverse Events (participants affected / at risk) | 97/104 | 92/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP101 (N=104) | Placebo (N=99)
Bronchitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pleurisy viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Traumatic hematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal hematoma (Renal and urinary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP101 (N=104) | Placebo (N=99)
Diarrhoea (Gastrointestinal disorders) | 57 | 50
Abdominal pain (Gastrointestinal disorders) | 36 | 60
Defaecation urgency (Gastrointestinal disorders) | 34 | 41
Abdominal distension (Gastrointestinal disorders) | 27 | 30
Nausea (Gastrointestinal disorders) | 28 | 28
Abdominal tenderness (Gastrointestinal disorders) | 22 | 31
Anal incontinence (Gastrointestinal disorders) | 19 | 22
Haematochezia (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 6 | 8
Constipation (Gastrointestinal disorders) | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 25 | 36
Dehydration (Metabolism and nutrition disorders) | 12 | 21
Urinary tract infection (Infections and infestations) | 7 | 7
Pyrexia (General disorders) | 7 | 11
Fatigue (General disorders) | 9 | 5
Pus in stool (Investigations) | 6 | 11
Headache (Nervous system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI are: (i) the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to eighteen months from the lock-down of all study data and (ii) the sponsor can require the removal of its confidential information from results communications and may delay release for a period of up to 60 days for the purpose of filing patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03110133/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03110133/SAP_001.pdf